CLINICAL TRIAL: NCT00260299
Title: Dietary Cholesterol and Defects in Cholesterol Synthesis in Mevalonate Kinase Deficiency
Status: Terminated | Type: Observational
Why Stopped: Not enough participants
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jean-Baptiste Roullet, Clinical Professor, Oregon Health and Science University
Other Study IDs: MKD dietary study
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Mevalonic Aciduria; Mevalonate Kinase Deficiency; Immune System Diseases; Periodic Fever Syndromes, Hereditary; Lipid Metabolism, Inborn Errors
Keywords: cholesterol defects; Mevalonic Aciduria; Mevalonate Kinase Deficiency; HIDS; Hyperimmunoglobulinemia with periodic fever syndrome; MKD; Lipid Metabolism, Inborn Errors; Periodic Fever Syndromes, hereditary; mevalonic acid; mevalonate kinase; cholesterol, dietary; Hyper IgD; Multiple malformations; Fever
MeSH Terms: conditions — Mevalonate Kinase Deficiency; Immune System Diseases; Hereditary Autoinflammatory Diseases; Lipid Metabolism, Inborn Errors; Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples, cells (fibroblasts) from skin biopsy tissue, DNA, urine and stool
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Participants wanted for study of mevalonate kinase deficiency (MKD), mevalonic aciduria, or hyperimmunoglobulinemia with periodic fever syndrome (HIDS).

Patients with MKD (mevalonic aciduria or hyperimmunoglobulinemia with periodic fever syndrome (HIDS)) may be eligible for a research study conducted at Oregon Health & Science University (OHSU) in Portland, Oregon USA. The purpose of the study is to find out more about how these diseases affect body chemistry and health. The researchers also want to find out how cholesterol in the diet affect blood cholesterol and how the body handles cholesterol. This is a short-term and long-term dietary study. The long-term goal of this research is to see if controlling dietary cholesterol can decrease any of the symptoms of the diseases.

The study could involve up to 12 one-week admissions to OHSU over the course of 5 years.

DETAILED DESCRIPTION:
Participants are admitted to the clinical research center for up to a week per visit. Additional visits at least yearly encouraged. During the week we measure such things as cholesterol absorption, sterol and bile acid synthesis, mevalonate and mevalonate shunt products, isoprenoids, fatty acids, leukotrienes, plasma cholesterol and other sterol levels. Also, the effects of altering dietary cholesterol on plasma 24-S OH-cholesterol, a measure of brain cholesterol turnover, will be evaluated. Studies of body composition/ metabolism/ growth, development, behavior, sleep, feeding, hearing and vision will be carried out to document the phenotype and determine if dietary intervention may be helpful.

The objective of the study is to characterize the metabolic and phenotypic consequences of MKD and study the effects of altering dietary cholesterol in MKD. We hypothesize that some of the phenotypic effects of MKD are due to altered cholesterol metabolism, but that the phenotype is predominantly due to derangements in isoprenoid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Must have documented mevalonate kinase deficiency, mevalonic aciduria, or HIDS
* Must be willing to participate in most research procedures

Exclusion Criteria:

* Unable or unwilling to participate in most research procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children or adults with mevalonic kinase deficiency/mevalonic aciduria/HIDS
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2005-02; Primary Completion 2014-12-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Determine the effects of dietary cholesterol changes in MKD on cholesterol and related synthetic pathways | December 2011
  blood levels of cholesterol

SECONDARY OUTCOMES:
Define genotype, phenotype and response to dietary cholesterol. Determine genotype-therapy correlations. | December 2011
  Gene Mutations - 7-dehydrocholesterol levels

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Steiner, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States